CLINICAL TRIAL: NCT04666298
Title: A Placebo-controlled, Double-blind, Randomized Trial to Evaluate the Effect of Different Doses of Inclisiran Given as Subcutaneous Injections in Japanese Participants With High Cardiovascular Risk and Elevated LDL-C
Brief Title: Study of Efficacy and Safety of Inclisiran in Japanese Participants With High Cardiovascular Risk and Elevated LDL-C
Acronym: ORION-15
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CKJX839A11201
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Results first posted 2023-05-10 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Hypercholesterolemia; Heterozygous Familial Hypercholesterolemia
Keywords: inclisiran; siRNA; dyslipidemia; PCSK9; Hypercholesterolemia; LDL-C
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 300 mg inclisiran sodium (Experimental): Subcutaneous injection
  Interventions: Drug: Inclisiran sodium
- 200 mg inclisiran sodium (Experimental): Subcutaneous injection
  Interventions: Drug: Inclisiran sodium
- 100 mg inclisiran sodium (Experimental): Subcutaneous injection
  Interventions: Drug: Inclisiran sodium
- Placebo (Placebo Comparator): Subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inclisiran sodium — Subcutaneously injected on Day 1, 90 and 270.
  Other Names: KJX839
  Arms: 100 mg inclisiran sodium; 200 mg inclisiran sodium; 300 mg inclisiran sodium
Drug: Placebo — Subcutaneously injected on Day 1, 90, and 270.
  Other Names: KJX839 placebo
  Arms: Placebo

SUMMARY:
This was a placebo-controlled, double-blind, randomized trial in Japanese participants with history of coronary artery disease (CAD) or participants categorized in 'high risk' by JAS 2017 guideline, or Japanese participants with heterozygous familial hypercholesterolemia (HeFH) and elevated Low-density lipoprotein cholesterol (LDL-C) despite maximum tolerated dose of statin(s) to evaluate the efficacy, safety, tolerability, and PK of subcutaneous inclisiran injection(s).

DETAILED DESCRIPTION:
The expected duration of the participants' involvement in the study was approximately 374 days which included screening (up to 14 days), Day 1 study drug administration, two additional injections on Day 90 and Day 270, and the follow-up period to Day 360.

The primary analysis was conducted after all participants had finished Day 180 visit assessments or discontinued before Day 180 visit.

After the primary analysis, double-blind treatment period were maintained to Day 360, although specific sponsor members (except for blinded monitors) were unblinded for the regulatory submission in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Participants with history of CAD or participants categorized in 'high risk' by Japan Atherosclerosis Society (JAS) 2017 guidelines or participants with heterozygous familial hypercholesterolemia (HeFH)
* As per the JAS 2017 guideline, participants not meeting the LDL-C management targets.
* Participants on statins should be receiving a maximally tolerated dose.
* Participants not receiving statins must have documented evidence of intolerance to at least one statin.
* The lipid-lowering therapy should have remained stable for ≥ 30 days before screening with no planned medication/ dose change until Day 180

Exclusion Criteria:

* Participants diagnosed with homozygous familial hypercholesterolemia (HoFH).
* Treatment (within 90 days of screening) with monoclonal antibodies directed towards PCSK9.
* New York Heart Association (NYHA) class IV heart failure or last known left ventricular ejection fraction <25%.
* Cardiac arrhythmia within 3 months prior to randomization that is not controlled by medication or via ablation.
* Uncontrolled hypertension: systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg prior to randomization despite antihypertensive therapy.
* Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver or unexplained elevations in alanine aminotransferase (ALT), aspartate aminotransferase (AST), >3x the upper limit of normal (ULN), or total bilirubin >2x ULN at screening.
* Severe concomitant non-cardiovascular disease that carries the risk of reducing life expectancy to less than 2 years.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (33):
- Japan (33):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Matsudo, Chiba
  - Novartis Investigative Site, Itoshima, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Nakagawa, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Sashima-gun, Ibaraki
  - Novartis Investigative Site, Tsuchiura, Ibaraki
  - Novartis Investigative Site, Kahoku-gun, Ishikawa-ken
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Komatsu, Ishikawa-ken
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Fujisawa, Kanagawa
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Kuse, Kyoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Ōmura, Nagasaki
  - Novartis Investigative Site, Izumisano, Osaka
  - Novartis Investigative Site, Matsubara, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Iruma-gun, Saitama
  - Novartis Investigative Site, Sayama, Saitama
  - Novartis Investigative Site, Chiyoda City, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Nerima-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Chuoh-ku
  - Novartis Investigative Site, Gifu
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Ōita
  - Novartis Investigative Site, Saga

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Warden BA, Duell PB. Inclisiran: A Novel Agent for Lowering Apolipoprotein B-containing Lipoproteins. J Cardiovasc Pharmacol. 2021 Aug 1;78(2):e157-e174. doi: 10.1097/FJC.0000000000001053. PMID 33990512
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1656

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo subcutaneous injection
- 100 mg Inclisiran Sodium: 100 mg inclisiran sodium (equivalent to 94.5 mg inclisiran) subcutaneous injection
- 200 mg Inclisiran Sodium: 200 mg inclisiran sodium (equivalent to 189 mg inclisiran) subcutaneous injection
- 300 mg Inclisiran Sodium: 300 mg inclisiran sodium (equivalent to 284 mg inclisiran) subcutaneous injection
Period: Overall Study
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Started | 57 | 55 | 101 | 99
Completed | 55 | 55 | 100 | 95
Not Completed | 2 | 0 | 1 | 4
Not completed — Subject decision | 1 | 0 | 0 | 2
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Protocol deviation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium | Total
Number analyzed (Participants) | 57 | 55 | 101 | 99 | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (11.12) | 62.7 (9.25) | 64.7 (10.57) | 63.0 (10.66) | 63.6 (10.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 21 | 22 | 80
  Male | 39 | 36 | 80 | 77 | 232
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 57 | 55 | 101 | 99 | 312

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) to Day 180
Description: Percent change from baseline in LDL-C was calculated to evaluate the effect of inclisiran at Day 180.
  Difference between different inclisiran dose groups and the placebo group in percentage change in LDL-C levels from baseline to Day 180 were calculated to capture both, the effect of the study drug and the effect of additional medications, mirroring the conditions in clinical practice.
  An MMRM (Mixed-effect Model with Repeated Measurement) was used as the primary analysis model, with treatment group, visits, interaction between visits and treatment groups, current use of statins or other lipid-modifying therapies as fixed effects, and baseline LDL-C as a continuous covariate.
Time Frame: Baseline, Day 180
Population: The FAS comprised all participants to whom study treatment had been assigned by randomization.
  The overall number of participants analyzed represents the participants in the Full Analysis Set (FAS) who had valid LDL-C value for both, baseline and day 180
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change in LDL-C
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Number analyzed (Participants) | 56 | 55 | 101 | 96
percent change in LDL-C | 9.0 [3.5 to 14.5] | -47.6 [-53.4 to -41.8] | -51.9 [-56.8 to -47.0] | -56.3 [-61.1 to -51.4]
Statistical Analysis 1: Comparison: Placebo vs 100 mg Inclisiran Sodium; Test type: Superiority; p < .0001, Mixed Models Analysis — One-sided adjusted p-value for multiple comparisons using Dunnett´s multiple t-test; Mean Difference (Net) = -56.6, 95% CI 2-sided [-64.2 to -49.0], Standard Error of Mean 3.24
Statistical Analysis 2: Comparison: Placebo vs 200 mg Inclisiran Sodium; Test type: Superiority; p < .0001, Mixed Models Analysis — One-sided adjusted p-value for multiple comparisons using Dunnett´s multiple t-test; Mean Difference (Net) = -60.9, 95% CI 2-sided [-67.6 to -54.3], Standard Error of Mean 2.84
Statistical Analysis 3: Comparison: Placebo vs 300 mg Inclisiran Sodium; Test type: Superiority; p < .0001, Mixed Models Analysis — One-sided adjusted p-value for multiple comparisons using Dunnett´s multiple t-test; Mean Difference (Net) = -65.3, 95% CI 2-sided [-72.0 to -58.6], Standard Error of Mean 2.86

2. Secondary Outcome: Percent Change From Baseline in PCSK9 by Visit
Description: Percent change from baseline in proprotein convertase subtilisin/kexin type 9 (PCSK9) was calculated to evaluate the effect of inclisiran over time.
Time Frame: Baseline, day 14, day 30, day 60, day 90, day 104, day 120, day 150, and day 180
Population: The overall number of participants analyzed represents the participants in the Full Analysis Set (FAS) who had at least one valid measurement of PCSK9.
  The number analyzed per row represents the participants with a valid PCSK9 value for both, baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: percent change in PCSK9
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Number analyzed (Participants) | 57 | 55 | 101 | 98
percent change in PCSK9
  Day 14 | 4.79 (21.623) | -55.42 (19.980) | -65.64 (13.677) | -69.56 (11.387)
  Day 30 | 1.92 (22.427) | -66.45 (12.341) | -72.94 (8.809) | -76.46 (8.561)
  Day 60 | -0.16 (22.656) | -62.56 (15.356) | -73.23 (10.692) | -76.52 (9.953)
  Day 90: number analyzed (Participants) | 57 | 55 | 101 | 97
  Day 90 | 2.12 (21.447) | -59.76 (14.503) | -70.49 (10.806) | -73.09 (11.525)
  Day 104: number analyzed (Participants) | 57 | 55 | 101 | 96
  Day 104 | 2.65 (28.624) | -69.05 (11.109) | -76.23 (9.017) | -78.55 (8.052)
  Day 120: number analyzed (Participants) | 55 | 55 | 101 | 95
  Day 120 | 0.99 (21.572) | -70.29 (11.543) | -77.03 (8.206) | -79.80 (6.994)
  Day 150: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 150 | 2.34 (23.353) | -66.02 (12.724) | -73.94 (17.139) | -77.12 (8.770)
  Day 180: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 180 | 2.78 (21.226) | -63.62 (14.012) | -70.99 (10.495) | -75.97 (9.885)

3. Secondary Outcome: Percent Change From Baseline in LDL-C by Visit
Description: Percent change from baseline in low-density lipoprotein cholesterol (LDL-C) was calculated to evaluate the effect of inclisiran over time.
Time Frame: Baseline, day 14, day 30, day 60, day 90, day 104, day 120 and day 150
Population: The overall number of participants analyzed represents the participants in the Full Analysis Set (FAS) who had at least one valid measurement of LDL-C.
  The number analyzed per row represents the participants with a valid LDL-C value for both, baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: percent change in LDL-C
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Number analyzed (Participants) | 57 | 55 | 101 | 98
percent change in LDL-C
  Day 14 | 1.68 (18.099) | -37.15 (21.855) | -42.08 (20.503) | -47.60 (19.889)
  Day 30 | 1.29 (13.068) | -52.20 (18.389) | -55.54 (17.501) | -62.77 (15.097)
  Day 60 | 0.24 (15.314) | -50.06 (19.173) | -55.61 (17.570) | -62.35 (13.976)
  Day 90: number analyzed (Participants) | 57 | 55 | 101 | 97
  Day 90 | 2.69 (14.332) | -46.39 (17.872) | -53.92 (17.186) | -61.51 (15.480)
  Day 104: number analyzed (Participants) | 57 | 55 | 101 | 96
  Day 104 | 1.20 (13.519) | -53.00 (19.001) | -60.33 (15.912) | -65.68 (15.321)
  Day 120: number analyzed (Participants) | 55 | 55 | 101 | 95
  Day 120 | 2.26 (14.854) | -54.91 (19.410) | -62.04 (16.742) | -67.23 (16.017)
  Day 150: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 150 | 4.27 (16.983) | -55.46 (18.817) | -60.55 (16.502) | -66.15 (15.197)

4. Secondary Outcome: Absolute Change in LDL-C From Baseline at Day 180
Description: Absolute change from baseline in low-density lipoprotein cholesterol (LDL-C) was calculated to evaluate the effect of inclisiran until Day 180.
Time Frame: Baseline, Day 180
Population: The overall number of participants analyzed represents the participants in the Full Analysis Set (FAS) who had valid LDL-C value for both, baseline and day 180
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Number analyzed (Participants) | 56 | 55 | 101 | 96
mg/dL | 13.2 [6.6 to 19.8] | -49.3 [-56.2 to -42.3] | -53.9 [-59.8 to -48.0] | -57.7 [-63.5 to -51.8]

5. Secondary Outcome: Proportion of Participants With LDL-C Greater Than 80% of Baseline Value at Day 180
Description: Proportion of participants with LDL-C greater than 80% of baseline value at Day 180 was calculated to evaluate the effect of inclisiran until Day 180.
  Subjects are counted if the LDL-C value is greater than '0.8*(LDL-C at Baseline - LDL-C at Day180) + LDL-C at Day180', or the LDL-C value is greater than or equal to the LDL-C at Baseline.
Time Frame: Baseline, Day 180
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Number analyzed (Participants) | 56 | 55 | 101 | 96
Participants | 35 | 0 | 0 | 0

6. Secondary Outcome: Proportion of Participants With Greater or Equal to 50% LDL-C Reduction From Baseline by Visit
Description: Proportion of participants with greater or equal to 50% LDL-C reduction from baseline was calculated to evaluate the effect of inclisiran over time.
Time Frame: Baseline, day 14, day 30, day 60, day 90, day 104, day 120, day 150, and day 180
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Number analyzed (Participants) | 57 | 55 | 101 | 98
Participants
  Day 14 | 1 | 17 | 40 | 45
  Day 30 | 0 | 31 | 63 | 83
  Day 60 | 0 | 26 | 64 | 75
  Day 90: number analyzed (Participants) | 57 | 55 | 101 | 97
  Day 90 | 0 | 22 | 58 | 76
  Day 104: number analyzed (Participants) | 57 | 55 | 101 | 96
  Day 104 | 0 | 32 | 77 | 82
  Day 120: number analyzed (Participants) | 55 | 55 | 101 | 95
  Day 120 | 0 | 37 | 72 | 82
  Day 150: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 150 | 0 | 35 | 73 | 78
  Day 180: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 180 | 0 | 33 | 68 | 73

7. Secondary Outcome: Percent Change From Baseline in Cholesterol by Visit
Description: Percent change from baseline in cholesterol by visit was calculated to evaluate the effect of inclisiran over time
Time Frame: Baseline, day 14, day 30, day 60, day 90, day 104, day 120, day 150, and day 180
Population: The overall number of participants analyzed represents the participants in the Full Analysis Set (FAS) who had at least one valid measurement of cholesterol.
  The number analyzed per row represents the participants with a valid cholesterol value for both, baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: Percent change in cholesterol
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Number analyzed (Participants) | 57 | 55 | 101 | 98
Percent change in cholesterol
  Day 14 | 0.87 (10.399) | -21.94 (14.034) | -24.71 (12.917) | -28.60 (12.476)
  Day 30 | 0.89 (9.003) | -30.92 (12.558) | -32.90 (11.739) | -37.09 (10.227)
  Day 60 | 0.31 (8.885) | -29.47 (13.426) | -33.71 (12.291) | -37.01 (9.948)
  Day 90: number analyzed (Participants) | 57 | 55 | 101 | 97
  Day 90 | 1.03 (8.952) | -27.30 (13.127) | -32.26 (12.103) | -36.34 (10.655)
  Day 104: number analyzed (Participants) | 57 | 55 | 101 | 96
  Day 104 | 1.62 (10.178) | -30.72 (13.239) | -35.63 (11.875) | -39.53 (10.468)
  Day 120: number analyzed (Participants) | 55 | 55 | 101 | 95
  Day 120 | 1.11 (10.860) | -32.24 (13.575) | -36.24 (12.995) | -39.38 (10.165)
  Day 150: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 150 | 2.41 (10.801) | -32.20 (14.246) | -35.70 (11.980) | -38.12 (10.850)
  Day 180: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 180 | 2.78 (10.272) | -30.22 (12.468) | -32.95 (12.540) | -35.46 (11.941)

8. Secondary Outcome: Percent Change From Baseline in Triglycerides by Visit
Description: Percent change from baseline in triglycerides by visit was calculated to evaluate the effect of inclisiran over time
Time Frame: Baseline, day 14, day 30, day 60, day 90, day 104, day 120, day 150, and day 180
Population: The overall number of participants analyzed represents the participants in the Full Analysis Set (FAS) who had at least one valid measurement of triglycerides.
  The number analyzed per row represents the participants with a valid triglycerides value for both, baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: percent change in triglycerides
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Number analyzed (Participants) | 57 | 55 | 101 | 98
percent change in triglycerides
  Day 14 | 5.49 (28.803) | 1.24 (29.630) | -1.16 (51.241) | -7.19 (23.817)
  Day 30 | 7.76 (35.248) | -4.72 (25.843) | -8.69 (25.450) | -8.37 (28.240)
  Day 60 | 9.68 (37.000) | -7.17 (28.427) | -9.26 (27.598) | -9.93 (26.405)
  Day 90: number analyzed (Participants) | 57 | 55 | 101 | 97
  Day 90 | 6.83 (33.204) | -1.87 (40.499) | -12.17 (26.204) | -9.99 (29.230)
  Day 104: number analyzed (Participants) | 57 | 55 | 101 | 96
  Day 104 | 11.86 (37.365) | -7.12 (26.145) | -5.81 (55.419) | -13.51 (26.915)
  Day 120: number analyzed (Participants) | 55 | 55 | 101 | 95
  Day 120 | 3.57 (33.870) | -9.40 (27.192) | -9.32 (33.471) | -12.33 (26.280)
  Day 150: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 150 | 3.33 (32.023) | -5.60 (42.988) | -12.65 (24.766) | -11.81 (28.623)
  Day 180: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 180 | -0.19 (32.161) | -2.34 (33.783) | -12.11 (39.414) | -13.67 (27.307)

9. Secondary Outcome: Percent Change From Baseline in HDL Cholesterol by Visit
Description: Percent change from baseline in high-density lipoprotein cholesterol (HDL-C) by visit was calculated to evaluate the effect of inclisiran over time
Time Frame: Baseline, day 14, day 30, day 60, day 90, day 104, day 120, day 150, and day 180
Population: The overall number of participants analyzed represents the participants in the Full Analysis Set (FAS) who had at least one valid measurement of HDL Cholesterol.
  The number analyzed per row represents the participants with a valid HDL Cholesterol value for both, baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: percent change in HDL Cholesterol
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Number analyzed (Participants) | 57 | 55 | 101 | 98
percent change in HDL Cholesterol
  Day 14 | 1.73 (8.765) | 3.00 (10.745) | 5.93 (12.164) | 4.38 (10.727)
  Day 30 | 1.94 (11.259) | 4.86 (10.450) | 9.89 (13.656) | 8.43 (12.740)
  Day 60 | 0.57 (10.677) | 6.80 (15.222) | 8.02 (15.411) | 9.15 (14.984)
  Day 90: number analyzed (Participants) | 57 | 55 | 101 | 97
  Day 90 | 0.56 (11.543) | 6.51 (16.297) | 10.86 (16.359) | 8.59 (16.546)
  Day 104: number analyzed (Participants) | 57 | 55 | 101 | 96
  Day 104 | 1.35 (14.817) | 8.69 (15.303) | 11.04 (16.443) | 8.99 (17.280)
  Day 120: number analyzed (Participants) | 55 | 55 | 101 | 95
  Day 120 | 4.20 (13.747) | 8.84 (13.432) | 12.65 (16.777) | 11.97 (18.300)
  Day 150: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 150 | 5.12 (13.587) | 7.51 (17.455) | 12.80 (16.337) | 11.68 (18.486)
  Day 180: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 180 | 8.25 (12.940) | 6.89 (17.051) | 15.95 (17.025) | 14.26 (20.158)

10. Secondary Outcome: Percent Change From Baseline in Non-HDL Cholesterol by Visit
Description: Percent change from baseline in non-HDL Cholesterol by visit was calculated to evaluate the effect of inclisiran over time
Time Frame: Baseline, day 14, day 30, day 60, day 90, day 104, day 120, day 150, and day 180
Population: The overall number of participants analyzed represents the participants in the Full Analysis Set (FAS) who had at least one valid measurement of non-HDL Cholesterol.
  The number analyzed per row represents the participants with a valid non-HDL Cholesterol value for both, baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: percent change in non-HDL Cholesterol
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Number analyzed (Participants) | 57 | 55 | 101 | 98
percent change in non-HDL Cholesterol
  Day 14 | 1.13 (13.511) | -31.37 (19.592) | -35.68 (18.056) | -41.16 (17.005)
  Day 30 | 1.03 (11.483) | -44.72 (16.270) | -47.99 (15.318) | -54.17 (12.815)
  Day 60 | 0.62 (11.841) | -43.39 (16.505) | -48.18 (15.146) | -54.10 (12.034)
  Day 90: number analyzed (Participants) | 57 | 55 | 101 | 97
  Day 90 | 1.75 (11.931) | -39.83 (16.485) | -47.20 (15.002) | -53.18 (13.236)
  Day 104: number analyzed (Participants) | 57 | 55 | 101 | 96
  Day 104 | 1.96 (12.067) | -46.10 (17.006) | -51.98 (14.344) | -57.74 (12.513)
  Day 120: number analyzed (Participants) | 55 | 55 | 101 | 95
  Day 120 | 0.82 (14.045) | -48.22 (17.301) | -53.52 (15.425) | -58.67 (12.175)
  Day 150: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 150 | 1.96 (13.519) | -47.90 (17.495) | -52.85 (14.254) | -56.82 (12.997)
  Day 180: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 180 | 1.29 (13.455) | -44.83 (15.558) | -50.15 (16.446) | -54.04 (14.230)

11. Secondary Outcome: Percent Change From Baseline in VLDL-C by Visit
Description: Percent change from baseline in very low-density lipoprotein cholesterol (VLDL - C) by visit was calculated to evaluate the effect of inclisiran over time
Time Frame: Baseline, day 14, day 30, day 60, day 90, day 104, day 120, day 150, and day 180
Population: The overall number of participants analyzed represents the participants in the Full Analysis Set (FAS) who had at least one valid measurement of VLDL-C.
  The number analyzed per row represents the participants with a valid VLDL-C value for both, baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: percent change in VLDL-C
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Number analyzed (Participants) | 57 | 55 | 101 | 98
percent change in VLDL-C
  Day 14 | 5.55 (28.428) | -2.96 (31.885) | -5.56 (43.055) | -12.41 (25.589)
  Day 30 | 6.69 (33.655) | -9.01 (28.560) | -13.39 (28.081) | -14.74 (30.582)
  Day 60 | 9.40 (36.824) | -10.27 (32.555) | -14.02 (28.944) | -17.94 (25.358)
  Day 90: number analyzed (Participants) | 57 | 55 | 101 | 97
  Day 90 | 6.53 (33.387) | -5.39 (41.490) | -16.70 (26.127) | -15.76 (27.957)
  Day 104: number analyzed (Participants) | 57 | 55 | 101 | 96
  Day 104 | 11.56 (37.588) | -12.10 (28.575) | -12.54 (45.978) | -24.05 (26.076)
  Day 120: number analyzed (Participants) | 55 | 55 | 101 | 95
  Day 120 | 3.10 (33.707) | -15.90 (30.271) | -14.05 (36.083) | -22.29 (24.030)
  Day 150: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 150 | 3.41 (31.791) | -10.91 (45.835) | -17.49 (27.270) | -18.39 (30.321)
  Day 180: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 180 | -0.30 (31.345) | -7.30 (33.946) | -17.89 (33.050) | -21.74 (27.746)

12. Secondary Outcome: Percent Change From Baseline in Apo- A1 by Visit
Description: Percent change from baseline in Apolipoprotein A1 (Apo-A1) by visit was calculated to evaluate the effect of inclisiran over time
Time Frame: Baseline, day 14, day 30, day 60, day 90, day 104, day 120, day 150, and day 180
Population: The overall number of participants analyzed represents the participants in the Full Analysis Set (FAS) who had at least one valid measurement of Apo-A1.
  The number analyzed per row represents the participants with a valid Apo-A1 value for both, baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: percent change in Apo-A1
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Number analyzed (Participants) | 57 | 55 | 101 | 98
percent change in Apo-A1
  Day 14 | 0.04 (8.872) | 3.64 (9.293) | 2.29 (7.659) | 3.98 (7.952)
  Day 30 | 0.90 (9.713) | 2.70 (10.553) | 4.52 (9.302) | 4.35 (9.012)
  Day 60 | 0.00 (8.501) | 4.71 (11.785) | 3.89 (10.196) | 5.18 (10.023)
  Day 90: number analyzed (Participants) | 57 | 55 | 101 | 97
  Day 90 | -0.35 (9.888) | 3.86 (11.353) | 5.71 (10.609) | 5.21 (10.383)
  Day 104: number analyzed (Participants) | 57 | 55 | 101 | 96
  Day 104 | 0.14 (10.780) | 5.89 (13.922) | 5.66 (11.007) | 4.99 (10.061)
  Day 120: number analyzed (Participants) | 55 | 55 | 101 | 95
  Day 120 | 1.79 (10.707) | 5.33 (12.293) | 6.49 (11.334) | 6.60 (11.152)
  Day 150: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 150 | 3.70 (11.571) | 4.85 (14.330) | 7.46 (11.582) | 8.35 (12.564)
  Day 180: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 180 | 6.09 (11.862) | 4.99 (14.170) | 10.26 (12.250) | 9.09 (13.871)

13. Secondary Outcome: Percent Change From Baseline in Apo- B by Visit
Description: Percent change from baseline in Apolipoprotein B (Apo-B) by visit was calculated to evaluate the effect of inclisiran over time
Time Frame: Baseline, day 14, day 30, day 60, day 90, day 104, day 120, day 150, and day 180
Population: The overall number of participants analyzed represents the participants in the Full Analysis Set (FAS) who had at least one valid measurement of Apo-B.
  The number analyzed per row represents the participants with a valid Apo-B value for both, baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: percent change in Apo-B
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Number analyzed (Participants) | 57 | 55 | 101 | 98
percent change in Apo-B
  Day 14 | 1.09 (13.795) | -28.16 (16.442) | -32.45 (17.518) | -37.12 (16.743)
  Day 30 | 2.16 (12.904) | -39.72 (14.749) | -43.99 (15.185) | -48.76 (12.962)
  Day 60 | 1.41 (11.965) | -39.94 (13.996) | -44.49 (14.654) | -48.53 (12.005)
  Day 90: number analyzed (Participants) | 57 | 55 | 101 | 97
  Day 90 | 2.76 (12.882) | -35.84 (14.134) | -42.04 (14.319) | -46.78 (12.611)
  Day 104: number analyzed (Participants) | 57 | 55 | 101 | 96
  Day 104 | 3.03 (13.304) | -40.86 (14.578) | -47.03 (13.283) | -51.93 (12.390)
  Day 120: number analyzed (Participants) | 55 | 55 | 101 | 95
  Day 120 | 2.05 (14.719) | -43.39 (14.174) | -48.18 (14.142) | -51.85 (12.414)
  Day 150: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 150 | 3.86 (13.559) | -42.82 (14.799) | -46.71 (13.775) | -50.41 (12.411)
  Day 180: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 180 | 3.82 (14.649) | -38.63 (13.265) | -44.50 (14.685) | -46.81 (13.968)

14. Secondary Outcome: Percent Change From Baseline in Lipoprotein-a by Visit
Description: Percent change from baseline in Lipoprotein a (LP(a)) by visit was calculated to evaluate the effect of inclisiran over time
Time Frame: Baseline, day 14, day 30, day 60, day 90, day 104, day 120, day 150, and day 180
Population: The overall number of participants analyzed represents the participants in the Full Analysis Set (FAS) who had at least one valid measurement of LP(a).
  The number analyzed per row represents the participants with a valid LP(a) value for both, baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: percent change in LP(a)
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Number analyzed (Participants) | 57 | 55 | 101 | 98
percent change in LP(a)
  Day 14 | 3.33 (32.912) | -21.77 (24.909) | -16.63 (41.372) | -22.84 (22.934)
  Day 30 | 0.92 (31.643) | -28.09 (21.846) | -22.80 (46.679) | -31.30 (26.785)
  Day 60 | -4.29 (30.944) | -30.89 (26.802) | -26.11 (45.964) | -36.21 (22.036)
  Day 90: number analyzed (Participants) | 57 | 55 | 101 | 97
  Day 90 | 4.35 (29.270) | -27.08 (25.260) | -24.93 (42.005) | -34.26 (25.027)
  Day 104: number analyzed (Participants) | 57 | 55 | 101 | 96
  Day 104 | -2.41 (26.326) | -32.02 (30.286) | -25.99 (45.444) | -37.92 (30.801)
  Day 120: number analyzed (Participants) | 55 | 55 | 101 | 95
  Day 120 | 0.22 (23.786) | -31.46 (27.979) | -30.26 (37.382) | -37.24 (25.389)
  Day 150: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 150 | 4.02 (32.703) | -32.21 (26.140) | -21.59 (47.820) | -38.11 (24.508)
  Day 180: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 180 | 5.45 (36.446) | -30.15 (25.578) | -25.46 (48.279) | -35.41 (25.123)

15. Secondary Outcome: Proportion of Participants Who Attain Lipid Control Target Pre-specified by JAS 2017 Guidelines for Their Level of Cardiovascular Risk at Day 180
Description: Proportion of participants who attain lipid control target pre-specified by Japan Atherosclerosis Society(JAS) 2017 guidelines for their level of cardiovascular risk at Day 180 was calculated to evaluate the effect of inclisiran.
Time Frame: Day 180
Population: The overall number of participants analyzed represents the participants in the Full Analysis Set (FAS) who had at least one valid measurement of LDL-C at Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Number analyzed (Participants) | 56 | 55 | 101 | 96
Participants | 5 | 50 | 87 | 91

16. Secondary Outcome: Number of Participants With LDL-C Levels of <25 mg/dL, <50 mg/dL, <70 mg/dL, and <100 mg/dL by Visit
Description: Number of participants by LDL-C levels was calculated to evaluate the effect of inclisiran.
Time Frame: Baseline, day 14, day 30, day 60, day 90, day 104, day 120, day 150, and day 180
Population: The overall number of participants analyzed represents the participants in the Full Analysis Set (FAS) who had at least one valid measurement of LDL-C.
  The number analyzed per row represents the participants with a valid LDL-C at that particular visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 100 mg Inclisiran Sodium | 200 mg Inclisiran Sodium | 300 mg Inclisiran Sodium
Number analyzed (Participants) | 57 | 55 | 101 | 98
Participants
  Day 14: LDL-C <25 mg/dL | 0 | 1 | 5 | 10
  Day 14: LDL-C <50 mg/dL | 1 | 19 | 38 | 43
  Day 14: LDL-C <70 mg/dL | 3 | 29 | 56 | 66
  Day 14: LDL-C <100 mg/dL | 22 | 45 | 81 | 86
  Day 30: LDL-C <25 mg/dL | 0 | 6 | 14 | 20
  Day 30: LDL-C <50 mg/dL | 0 | 30 | 56 | 71
  Day 30: LDL-C <70 mg/dL | 3 | 40 | 74 | 80
  Day 30: LDL-C <100 mg/dL | 22 | 51 | 93 | 94
  Day 60: LDL-C <25 mg/dL | 0 | 6 | 14 | 23
  Day 60: LDL-C <50 mg/dL | 0 | 28 | 57 | 70
  Day 60: LDL-C <70 mg/dL | 5 | 37 | 77 | 79
  Day 60: LDL-C <100 mg/dL | 21 | 50 | 92 | 92
  Day 90: LDL-C <25 mg/dL: number analyzed (Participants) | 57 | 55 | 101 | 97
  Day 90: LDL-C <25 mg/dL | 0 | 2 | 12 | 21
  Day 90: LDL-C <50 mg/dL: number analyzed (Participants) | 57 | 55 | 101 | 97
  Day 90: LDL-C <50 mg/dL | 0 | 27 | 51 | 67
  Day 90: LDL-C <70 mg/dL: number analyzed (Participants) | 57 | 55 | 101 | 97
  Day 90: LDL-C <70 mg/dL | 1 | 35 | 74 | 80
  Day 90: LDL-C <100 mg/dL: number analyzed (Participants) | 57 | 55 | 101 | 97
  Day 90: LDL-C <100 mg/dL | 24 | 49 | 93 | 94
  Day 104: LDL-C <25 mg/dL: number analyzed (Participants) | 57 | 55 | 101 | 96
  Day 104: LDL-C <25 mg/dL | 0 | 6 | 22 | 27
  Day 104: LDL-C <50 mg/dL: number analyzed (Participants) | 57 | 55 | 101 | 96
  Day 104: LDL-C <50 mg/dL | 0 | 30 | 64 | 70
  Day 104: LDL-C <70 mg/dL: number analyzed (Participants) | 57 | 55 | 101 | 96
  Day 104: LDL-C <70 mg/dL | 4 | 38 | 82 | 80
  Day 104: LDL-C <100 mg/dL: number analyzed (Participants) | 57 | 55 | 101 | 96
  Day 104: LDL-C <100 mg/dL | 25 | 52 | 95 | 92
  Day 120: LDL-C <25 mg/dL: number analyzed (Participants) | 55 | 55 | 101 | 95
  Day 120: LDL-C <25 mg/dL | 0 | 9 | 25 | 32
  Day 120: LDL-C <50 mg/dL: number analyzed (Participants) | 55 | 55 | 101 | 95
  Day 120: LDL-C <50 mg/dL | 0 | 32 | 64 | 70
  Day 120: LDL-C <70 mg/dL: number analyzed (Participants) | 55 | 55 | 101 | 95
  Day 120: LDL-C <70 mg/dL | 3 | 39 | 82 | 81
  Day 120: LDL-C <100 mg/dL: number analyzed (Participants) | 55 | 55 | 101 | 95
  Day 120: LDL-C <100 mg/dL | 24 | 53 | 95 | 91
  Day 150: LDL-C <25 mg/dL: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 150: LDL-C <25 mg/dL | 0 | 5 | 24 | 31
  Day 150: LDL-C <50 mg/dL: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 150: LDL-C <50 mg/dL | 0 | 32 | 67 | 71
  Day 150: LDL-C <70 mg/dL: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 150: LDL-C <70 mg/dL | 2 | 41 | 81 | 81
  Day 150: LDL-C <100 mg/dL: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 150: LDL-C <100 mg/dL | 23 | 52 | 95 | 93
  Day 180: LDL-C <25 mg/dL: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 180: LDL-C <25 mg/dL | 0 | 7 | 13 | 26
  Day 180: LDL-C <50 mg/dL: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 180: LDL-C <50 mg/dL | 0 | 30 | 56 | 65
  Day 180: LDL-C <70 mg/dL: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 180: LDL-C <70 mg/dL | 2 | 40 | 78 | 80
  Day 180: LDL-C <100 mg/dL: number analyzed (Participants) | 56 | 55 | 101 | 96
  Day 180: LDL-C <100 mg/dL | 22 | 54 | 94 | 90

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment up to a maximum duration of 360 days
Groups:
- Inclisiran 100 mg: 100 mg inclisiran sodium (equivalent to 94.5 mg inclisiran) subcutaneous injection
- Inclisiran 200 mg: 200 mg inclisiran sodium (equivalent to 189 mg inclisiran) subcutaneous injection
- Inclisiran 300 mg: 300 mg inclisiran sodium (equivalent to 284 mg inclisiran) subcutaneous injection
Arm/Group | Placebo | Inclisiran 100 mg | Inclisiran 200 mg | Inclisiran 300 mg
All-Cause Mortality (participants affected / at risk) | 1/57 | 0/55 | 0/101 | 0/99
Serious Adverse Events (participants affected / at risk) | 6/57 | 2/55 | 7/101 | 7/99
Other Adverse Events (participants affected / at risk) | 32/57 | 38/55 | 59/101 | 59/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=57) | Inclisiran 100 mg (N=55) | Inclisiran 200 mg (N=101) | Inclisiran 300 mg (N=99)
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Epiretinal membrane (Eye disorders) | 0 | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 1 | 0 | 0 | 0
Vascular stent stenosis (General disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Embolic cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=57) | Inclisiran 100 mg (N=55) | Inclisiran 200 mg (N=101) | Inclisiran 300 mg (N=99)
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 5 | 1
Injection site reaction (General disorders) | 2 | 3 | 12 | 6
Malaise (General disorders) | 6 | 1 | 2 | 7
Pyrexia (General disorders) | 7 | 8 | 12 | 18
Vaccination site pain (General disorders) | 8 | 1 | 5 | 5
COVID-19 (Infections and infestations) | 2 | 8 | 5 | 6
Herpes zoster (Infections and infestations) | 3 | 1 | 3 | 0
Nasopharyngitis (Infections and infestations) | 3 | 4 | 6 | 7
Contusion (Injury, poisoning and procedural complications) | 3 | 4 | 3 | 3
Blood creatine phosphokinase increased (Investigations) | 4 | 1 | 3 | 5
C-reactive protein increased (Investigations) | 0 | 1 | 1 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 11 | 12 | 12
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 9 | 7 | 10 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 6 | 3 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 5
Headache (Nervous system disorders) | 5 | 3 | 3 | 3
Hypoaesthesia (Nervous system disorders) | 4 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT04666298/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT04666298/SAP_001.pdf